CLINICAL TRIAL: NCT00964093
Title: The Efficacy of Silver Alginate (Algidex®) Dressing in Reducing Central Line Infections in Very Low Birth Weight (VLBW) Infants: A Multicenter Collaborative Randomized Controlled Trial.
Brief Title: The Effectiveness of Silver Alginate (Algidex) Patch in the Prevention of Central Line Infections in Very Low Birth Weight Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Baylor Research Institute (Other)
Collaborators: DeRoyal Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Baylor IRB # 008-299
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Central Line Bloodstream Infections
Keywords: premature; infection; central line; very low birth weight; silver alginate; Algidex; neonatal; NICU
MeSH Terms: conditions — Premature Birth; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- No intervention (No Intervention)
  Interventions: Device: Silver Alginate

INTERVENTIONS:
Device: Silver Alginate — (Algidex ™)

SUMMARY:
The purpose of this study is to determine whether silver alginate (Algidex) patch is effective in the prevention of central line infections in very low birth weight infants.

DETAILED DESCRIPTION:
With rapid technological advancement, the increased use of vascular catheters has not only improved patient care strategies, but also contributed to the risk of infection. Unfortunately, catheter related blood stream infections still remain one of the major causes of morbidity in VLBW infants. In the United States, approximately 850,000 infections are attributed to catheters annually, occurring primarily in intensive care unit patients. The National Institute of Child Health and Human Development stated that 20% of infants less than 1500 grams will have at least one positive blood culture delaying their stay in the neonatal intensive care unit (NICU).

One approach to reducing the incidence of infection could be utilizing the antimicrobial properties of silver. Silver alginate has been proven safe and beneficial in the adult population in preventing catheter related infections. Studies done in mice and rats suggest acute toxicity occurring when the animals were given 23 mg of silver acetate/kg of body weight and chronic toxicity noticed when animals were given 1.5 mg/kg/day (5) Chronic toxicity in humans was shown with ingestion of 13 mg/kg/day (3) In our recently concluded pilot randomized controlled trial done in VLBW infants, safety of silver alginate was demonstrated by lack of skin reactions to the patches and mild increase in serum silver level ( Khattak et al; Pediatrics research March 2008, clinicaltrials.gov id: NCT00593684 ). However, there is no clinical evidence of efficacy in VLBW neonatal population. Based on the data from our pilot safety study, we hypothesize that using silver alginate dressing in this population will be efficacious in the prevention of blood stream infections. Although initial studies suggest that absorbed silver is not in a range toxic to human infants, we will continue to monitor silver levels in certain infants.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with birth weights between 500 and 1500 grams admitted to the NICU with any of the following lines will be eligible for inclusion in this study

   1. umbilical arterial line (UAL)
   2. umbilical venous line (UVL)
   3. peripheral arterial line (PAL)
   4. peripheral long line (PLL)
   5. central venous line (CVL)
2. Each eligible subject will be randomized to receive either standard of care or silver alginate dressing. Dressings will be changed every 7 days in accordance to current facility protocols.

Exclusion Criteria:

1. Any infant born with a lethal abnormality or who has received topical Silver therapy will be excluded from the study.

Ages: 1 Day to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2009-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this trial is to assess the efficacy of silver alginate dressing in reducing central line infections in VLBW infants | 2 years

SECONDARY OUTCOMES:
The secondary objectives are to compare mortality and total days of hospitalization between the groups. Safety will be assessed by obtaining silver levels, skin integrity, and adverse events related to the dressing. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Asif Khattak, MD, Principal Investigator — Baylor Health Care System; David M Kanter, MD, Principal Investigator — St. Mary's Medical Center, West Palm Beach, FL
Locations (1):
- Baylor University Medical Center - Women and Children's Services, Dallas, Texas, United States